CLINICAL TRIAL: NCT01450423
Title: Physical Exercise in Subjects With Juvenile Myoclonic Epilepsy Aged 15-50: A Randomized Controlled Trial
Brief Title: Physical Exercise in Subjects With Juvenile Myoclonic Epilepsy
Acronym: EFA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lars Bo Andersen (Other)
Responsible Party: Sponsor-Investigator, Lars Bo Andersen, Professor, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-20110080
Record Dates: First submitted 2011-10-09; First posted 2011-10-12 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Epilepsy; Epilepsia; Epileptic Seizures; Seizure Disorder
Keywords: Epilepsy; Physical activity; Cardio exercise; Physical fitness; Cognitive function
MeSH Terms: conditions — Epilepsy; Seizures; Motor Activity | interventions — Exercise

ARMS (2):
- Physical activity (Experimental)
  Interventions: Behavioral: Physical activity
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Physical activity — Participation in a 10-week supervised cardio exercise program two-three times a week. Each training session consists of 10 minutes of warm-up, 20 minutes treadmill run/walk and 30 minutes cycling. Heart rate (HR) is monitored during each session. Week 1-5: at least 15 minutes above 75% of HRmax in each session. Week 6-10: at least one session above 75% HRmax.
  Other Names: Cardio exercise program; Cardio training program
  Arms: Physical activity

SUMMARY:
Epilepsy is a chronic neurologic disorder characterized by seizures. Beside seizures people suffering from epilepsy experience several challenges related to education, work and everyday life such as learning-, problem-solving-, memory-, concentration-, attention difficulties and fatigue.

It is generally approved that physical activity (PA) has a positive effect on physical as well as mental factors. However, people with epilepsy are found to be less active and PA is rarely offered or recommended as supplement to anti-epileptic medical treatment. Few studies have investigated the effect of PA in subjects with epilepsy and additional studies of high methodical quality are needed to enable evidence-based information and counselling.

This study is carried through as a randomized controlled trial which investigates the effect of participation in a 10-week cardio exercise program in people with Juvenile Myoclonic Epilepsy aged 15-50.

The study hypothesis is that participation in a 10-week cardio exercise program will induce a positive change in cognitive function (concentration and attention) and possibly in brain-derived neurotrophic factor (BDNF). In addition it is expected that the intensity and duration of the 10-week cardio exercise program is sufficient to cause changes in physiological parameters related to a reduced risk of lifestyle diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age: 15-50
* Resident: Fyen, Denmark
* Epileptic syndrome: Juvenile Myoclonic Epilepsy

Exclusion Criteria:

* Physical handicaps which complicate participation in physical activity

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Cognitive function (concentration and attention) | Before and after a 10-week intervention period
  To assess cognitive function the following tests are used: Connor's Continuous Performance Test (CPT II), Trail Making Test part A and part B, Digit Symbol Modalities Test
physical fitness | Before and after a 10-week intervention period
  To assess physical fitness the following test are used: Wattmax test

SECONDARY OUTCOMES:
Brain-derived neurotrophic factor (BDNF) | Before and after a 10-week intervention period (chronic and acute)
  The chronic level of serum brain-derived neurotrophic factor (BDNF) is assessed in fasting blood samples. The acute level of serum BDNF is assessed in blood samples drawn immediately after completed wattmax test.
Bone mineral density | Before and after a 10-week intervention period
  To assess bone mineral density the following test is used: DEXA-scanning
Thyroidea Stimulating Hormone (TSH) | Before and after a 10-week intervention period
  The level of serum Thyroidea Stimulating Hormone (TSH) is assessed in fasting blood samples.
Insulin | Before and after a 10-week intervention period
  The level of insulin is assessed in fasting blood samples.
Glucose | Before and after a 10-week intervention period
  The level of glucose is assessed in fasting blood samples
Lipids | Before and after a 10-week intervention period
  The levels of lipids are assessed in fasting blood samples.
C-reactive-protein | Before and after a 10-week intervention period
  The level of c-reactive-protein is assessed in fasting blood samples.
Seizure frequency | Before and after a 10-week intervention period
  Seizure frequency is assessed by a neurologist using a standard seizure calender.
Blood pressure | Before and after a 10-week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bo Andersen, Professor, Principal Investigator — Center of Research in Childhood Health (RICH), University of Southern Denmark
Locations (2):
- Denmark (2):
  - Center of Research in Childhood Health, University of Southern Denmark, Odense, Region Syddanmark
  - Epilepsy clinic, Odense University Hospital, Odense, Region Syddanmark

REFERENCES:
- See also: Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark — http://www.sdu.dk/om_sdu/institutter_centre/iob_idraet_og_biomekanik